CLINICAL TRIAL: NCT02720822
Title: A Pragmatic, Phase III, Multi-site, Double-blind, Placebo Controlled, Parallel Arm, Dose Increment Randomised Trial of Regular, Low Dose Extended Release Morphine for Chronic Refractory Breathlessness
Brief Title: Breathlessness Exertion and Morphine Sulphate
Acronym: BEAMS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Flinders University (Other)
Responsible Party: Principal Investigator, David Currow, Professor: Palliative and Supportive Services, Flinders University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 030/15
Record Dates: First submitted 2016-03-10; First posted 2016-03-28 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Chronic Obstructive Pulmonary Disease; Dyspnea
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Morphine; Laxatives; Dioctyl Sulfosuccinic Acid; Sennosides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (12):
- Placebo (Placebo Comparator): Double-blind placebo capsule, looking identical to capsules with active treatment, during all three treatment weeks.
  Interventions: Drug: Placebo; Drug: Plus placebo laxative; Device: FitBit charge HR (Accelerometer)
- Morphine Sulfate (0, 0, 8 mg) (Experimental): Placebo on weeks one and two. Morphine 8 mg/day on week three.
  Interventions: Drug: Placebo; Drug: Morphine Sulfate; Drug: Plus laxative (Docusate with senna); Drug: Plus placebo laxative; Device: FitBit charge HR (Accelerometer)
- Morphine sulfate (0, 8, 8 mg) (Experimental): Placebo on week one. Morphine 8 mg/day on weeks two and three.
  Interventions: Drug: Placebo; Drug: Morphine Sulfate; Drug: Plus laxative (Docusate with senna); Drug: Plus placebo laxative; Device: FitBit charge HR (Accelerometer)
- Morphine sulfate (0, 8, 16 mg) (Experimental): Placebo on week one. Morphine 8 mg/day on week two. Morphine 16 mg/day on week three.
  Interventions: Drug: Placebo; Drug: Morphine Sulfate; Drug: Plus laxative (Docusate with senna); Drug: Plus placebo laxative; Device: FitBit charge HR (Accelerometer)
- Morphine sulfate (8, 8, 8 mg) (Experimental): Morphine 8 mg/day on weeks one, two and three.
  Interventions: Drug: Morphine Sulfate; Drug: Plus laxative (Docusate with senna); Device: FitBit charge HR (Accelerometer)
- Morphine sulfate (8, 8, 16 mg) (Experimental): Morphine 8 mg/day on weeks one and two. Morphine 16 mg/day on week three.
  Interventions: Drug: Morphine Sulfate; Drug: Plus laxative (Docusate with senna); Device: FitBit charge HR (Accelerometer)
- Morphine sulfate (8, 16, 16 mg) (Experimental): Morphine 8 mg/day on week one. Morphine 16 mg/day on weeks two and three.
  Interventions: Drug: Morphine Sulfate; Drug: Plus laxative (Docusate with senna); Device: FitBit charge HR (Accelerometer)
- Morphine sulfate (8, 16, 24 mg) (Experimental): Morphine 8 mg/day on week one. Morphine 16 mg/day on week two. Morphine 24 mg/day on week three.
  Interventions: Drug: Morphine Sulfate; Drug: Plus laxative (Docusate with senna); Device: FitBit charge HR (Accelerometer)
- Morphine sulfate (16, 16, 16 mg) (Experimental): Morphine 16 mg/day on weeks one, two and three.
  Interventions: Drug: Morphine Sulfate; Drug: Plus laxative (Docusate with senna); Device: FitBit charge HR (Accelerometer)
- Morphine sulfate (16, 16, 24 mg) (Experimental): Morphine 16 mg/day on weeks one and two. Morphine 24 mg/day on week three.
  Interventions: Drug: Morphine Sulfate; Drug: Plus laxative (Docusate with senna); Device: FitBit charge HR (Accelerometer)
- Morphine sulfate (16, 24, 24 mg) (Experimental): Morphine 16 mg/day on week one. Morphine 24 mg/day on weeks two and three.
  Interventions: Drug: Morphine Sulfate; Drug: Plus laxative (Docusate with senna); Device: FitBit charge HR (Accelerometer)
- Morphine sulfate (16, 24, 32 mg) (Experimental): Morphine 16 mg/day on week one. Morphine 24 mg/day on week two. Morphine 32 mg/day on week three.
  Interventions: Drug: Morphine Sulfate; Drug: Plus laxative (Docusate with senna); Device: FitBit charge HR (Accelerometer)

INTERVENTIONS:
Drug: Placebo — Treatment with placebo is given as one double-blind capsule in the morning.
  Other Names: MP342
  Arms: Morphine Sulfate (0, 0, 8 mg); Morphine sulfate (0, 8, 16 mg); Morphine sulfate (0, 8, 8 mg); Placebo
Drug: Morphine Sulfate — Treatment with sustained-release morphine sulfate is given as one double-blind capsule in the morning.
  Other Names: Kapanol (R)
  Arms: Morphine Sulfate (0, 0, 8 mg); Morphine sulfate (0, 8, 16 mg); Morphine sulfate (0, 8, 8 mg); Morphine sulfate (16, 16, 16 mg); Morphine sulfate (16, 16, 24 mg); Morphine sulfate (16, 24, 24 mg); Morphine sulfate (16, 24, 32 mg); Morphine sulfate (8, 16, 16 mg); Morphine sulfate (8, 16, 24 mg); Morphine sulfate (8, 8, 16 mg); Morphine sulfate (8, 8, 8 mg)
Drug: Plus laxative (Docusate with senna) — If patients are taking morphine, a laxative will be offered. This applies whatever the dose of morphine being taken (8mg, 16mg, 24mg or 32 mg).
  Arms: Morphine Sulfate (0, 0, 8 mg); Morphine sulfate (0, 8, 16 mg); Morphine sulfate (0, 8, 8 mg); Morphine sulfate (16, 16, 16 mg); Morphine sulfate (16, 16, 24 mg); Morphine sulfate (16, 24, 24 mg); Morphine sulfate (16, 24, 32 mg); Morphine sulfate (8, 16, 16 mg); Morphine sulfate (8, 16, 24 mg); Morphine sulfate (8, 8, 16 mg); Morphine sulfate (8, 8, 8 mg)
Drug: Plus placebo laxative — If the patients are taking placebo, a placebo laxative will be offered.
  Arms: Morphine Sulfate (0, 0, 8 mg); Morphine sulfate (0, 8, 16 mg); Morphine sulfate (0, 8, 8 mg); Placebo
Device: FitBit charge HR (Accelerometer) — A Fitbit will be worn by patients during week 1 and week 3.

SUMMARY:
Breathlessness is an overwhelming symptom affecting tens of thousands of Australians every day. For many people, it persists even when all the underlying causes have been optimally managed (chronic breathlessness). In these circumstances, it often occurs at rest or with minimal exertion.

Evidence from a number of clinical studies suggests that a small, regular dose of morphine helps to reduce safely the sensation of breathlessness. However, it is not well established which patients derive more benefit and what is the net clinical effect of this treatment (weighing benefits and harms).

This is a phase III, multi-site, randomised, double-blind, placebo-controlled trial with patients with chronic obstructive pulmonary disease (COPD) and severe chronic breathlessness which will explore several important questions:

* Are regular, low doses of morphine at four possible doses over 3 weeks more effective than placebo at improving breathlessness?
* Does increasing the dose in people who already are experiencing some benefit provide even greater reduction in worst breathlessness?
* Does the medication have any effect on daily activity and quality of life?
* What are the common or serious side effects of this intervention?
* Does the benefit from the medication outweigh the side effects it produces?
* Are there specific characteristics of people who are more likely to receive benefit from extended release morphine?

Participants will receive once daily extended release morphine (plus laxative, docusate with senna), or placebo (placebo laxative) in addition to their usual medication for up to 3 weeks at increasing doses.

Participants will have a medical interview and physical examination to collect some general health information, and baseline measurements including; daily activity, symptoms, and quality of life. A small amount of blood may be required to check eligibility. Further blood samples may be taken at week 1 and 3 to enable testing on how individuals respond to opioids, further consent will be obtained for these samples.

Data on benefits, side effects, and medical care will be collected during comprehensive weekly visits. Participants will also fill out a simple diary twice daily for weeks one to three of the study, and for one day each week during an optional 6 month extension stage.

The outcome of this study may enable better management of symptoms and activity in people COPD with medicines that are shown to be effective and safe.

DETAILED DESCRIPTION:
Background: Three hundred thousand (300,000) Australians are breathless at rest or on minimal exertion, often for years, despite optimal treatment of the underlying cause(s). This includes more than 70,000 people who are too breathless to leave their homes often for long periods of time. Underlying causes for such severe and ongoing breathlessness include chronic obstructive pulmonary disease (COPD), interstitial lung disease, heart failure, neurodegenerative diseases such as motor neurone disease and cachexia from any cause. The prevalence of chronic refractory breathlessness will continue to increase as the population ages because the chronic progressive diseases where breathlessness is common are increasing in prevalence. Nearly one half of all people experience distressing breathlessness during the last year of life.

The American Thoracic Society defines breathlessness as "a subjective experience of breathing discomfort that consists of qualitatively distinct sensations that vary in intensity".

Internationally, no medication is registered for the symptomatic reduction of chronic refractory breathlessness despite recommendations from the American Thoracic Society, the American College of Physicians, the Canadian Thoracic Society and the American College of Chest Physicians that regular, low-dose morphine is the evidence-based pharmaceutical option.

Aim: To enhance the evidence base for the pharmacological treatment of chronic refractory breathlessness using potential therapies compared to placebo.

Primary objective: To compare the difference of the net clinical effect (benefits and harms) on chronic refractory breathlessness in people with chronic obstructive pulmonary disease (COPD) and baseline breathlessness of 3 or 4 on the modified Medical Research Council breathlessness scale (mMRC) taking once daily, extended release oral morphine at two different doses when compared to placebo.

Co-primary objective: To compare the difference in steps per day measured using the FitbitR between people taking once daily, extended release oral morphine , by dosing level.

Secondary objectives

1. Is regular, low dose extended release oral morphine safe, including when the dose is titrated upwards, in a population of people with refractory breathlessness and COPD?
2. Do people whose breathlessness is helped by regular, low dose extended release oral morphine get additional benefit by further increasing the dose of morphine?
3. Over what period of time does benefit continue to increase once a dose level with benefit is achieved?
4. What percentage of people derive clinically significant benefit at each of four dosing levels, over and above placebo?
5. At the lower doses, is there evidence that any benefit does not last the full 24 hours? (end-of-dose failure)
6. Can we predict response, benefit and side effects from baseline demographic and clinical data in those people who get morphine?
7. Does the treatment of breathlessness with regular, low dose morphine have any effect on general health status and quality of life?
8. Is there any difference in activities of daily living in those treated with regular, low dose extended release oral morphine when compared to placebo.
9. Assess any effects of each treatment on anxiety and depression.
10. Understand the longer term benefits and side effects from extended release morphine in people with COPD when compared to placebo.
11. Do participants, while still blinded, have any preference at the end of the three week study?
12. Do caregivers notice any change in the burden and challenge of caregiving if the person they care for receives regular, low dose, extended release oral morphine for chronic breathlessness?
13. Do participants experience withdrawal from opioids at the end of the study as study medication ceases?

Sub-studies

1. Identify pharmacokinetic and pharmacodynamic parameters that may help to predict which individuals will achieve the greatest benefit in week one of therapy (8mg/day, 16mg/day).
2. Identify pharmacogenomic variations in opioid receptors and signaling that may help to predict clinical response (benefit, side effects or no response).
3. Study the effect on sleep in people participating in the study
4. Compare the impact on simulated driving in a sub-group of participants using commercially available driving simulators
5. Compare caregiver self-efficacy at the end of weeks one and three between groups when compared to baseline.
6. Compare the within trial incremental cost and cost effectiveness of the therapy
7. Evaluate any changes in total testosterone from baseline to the end of the 6-month extension.

Null hypothesis #1: In people who have COPD with refractory breathlessness, there is no difference in worst breathlessness intensity in the previous 24 hours with the addition of regular, low dose oral extended release morphine when compared to placebo.

Alternative hypothesis #1: The addition of regular, low dose oral extended release morphine reduces the intensity of worst breathlessness in the previous 24 hours in people with COPD and chronic breathlessness.

Null hypothesis #2: In people who have COPD with refractory breathlessness, there is no difference in the number of steps taken each day with the addition of regular, low dose oral extended release morphine when compared to placebo.

Alternative hypothesis #2: The addition of regular, low dose oral extended release morphine increases people's activities in people with COPD and chronic breathlessness.

Study design:

A five stage, national, multi-site, double-blind, parallel arm, block randomised, placebo controlled, factorial, dose increment phase III study of opioids for chronic refractory breathlessness in people with COPD:

Stage 0 - baseline (2 days); Stage 1 - randomisation #1 (1 week); Stage 2 - randomisation #2 (1 week); Stage 3 - randomisation #3 (1 week); and Stage 4 - an optional blinded extension arm (up to 6 months).

Stage 0. Baseline assessment: All consenting participants will complete 2 full days of baseline diary (evening) in order to become accustomed to completing the diary regularly and to provide stable baseline data regarding breathlessness, symptoms and activity (as measured by FitBit®). At completion of the 2 days, the participant will be reviewed, complete the remaining baseline assessments (questionnaires, measures and baseline safety data), and will then be eligible to be randomised the first time.

Time period: Two full days (4 diary entries)

Stage 1. Randomisation #1: Randomisation to mane orally: placebo OR 8mg extended release morphine OR 16mg extended release morphine. Daily diary. A FitBit will be worn this week. Participants randomised to extended release morphine will also receive blinded docusate with sennosides, while those randomised to placebo will receive identical laxative placebo. This is the primary outcome (end point) of the study.

Time period: 1 week

Stage 2. Randomisation #2: While continuing the arm assigned in Stage 1, add a randomisation to mane orally: placebo OR 8mg extended release morphine. Daily diary. Participants who were randomised to placebo in Stage 1 and extended release morphine in Stage 2 will have blinded docusate with sennosides replace the laxative placebo.

Time period: 1 week

Stage 3. Randomisation #3: While continuing the arm assigned in Stages 1 and 2, add a third randomisation to mane orally: placebo OR 8mg extended release morphine. Daily diary. A FitBit will be worn this week. Participants who were randomised to placebo in Stages 1 and 2 and extended release morphine in Stage 3 will have blinded docusate with sennosides replace the laxative placebo.

Time period: 1 week

Stage 4. Extension (optional for each individual participant): Continue double blind medications from Stages 1, 2 and 3 for up to six months. Diary one day each week. A blood test at the end of the six months will be taken for total testosterone levels.

Time period: up to 6 months.

Target population: This study is for people with optimally treated chronic breathlessness (modified Medical Research Council Scale (mMRC) of 3 or 4) and chronic obstructive pulmonary disease (COPD).

Primary outcome and its assessment: Change in the worst intensity of breathlessness in the previous 24 hours each morning, measured using an 11 point Numerical Rating Scale, recorded in the evening diary entry by participants.

Significance: The study will answer several practical questions including whether regular, low dose extended release oral morphine delivers a net benefit in people with COPD in reducing breathlessness on exertion (worst breathlessness in a 24 hour period) in steady state; whether dose increases beyond initial response provide a greater net benefit; the pattern of symptomatic response in the days after successful titration; and the proportion of people who derive a clinically meaningful symptomatic benefit at each dose level.

Analysis plan: All analyses will be conducted on an intention-to-treat basis. Missing data will be imputed using multiple imputation with 50 resamples drawn. The primary comparisons on which the study is powered are at the end of week 1: placebo compared to 8mg extended release morphine daily; and placebo compared to 16mg extended release morphine daily. Change in breathlessness in the first week between these groups will be evaluated using a random effects mixed model.

Sample size calculation All calculations assume Type I (family wise error rate (FWER)) error rate of 5% and Type II error rate of 20% (power of 80%) respectively. The primary analyses comprise two comparisons made at the end of week 1 (placebo compared to 8mg and placebo compared to 16mg), each assessed at alpha = 0.025 (two-sided) to protect the overall type 1 error rate. Using the variance-covariance matrix and mean responses from data arising from the MOP study, it was found through simulations (n = 1000) and using a mixed model analysis over 8 days, that 45 subjects per group are required to detect a difference of 1.09 NRS units where the standard deviation at each day varied between 2.0 and 2.5 NRS units.

The second family comprises one comparison, involving only those subjects who improved by 1.09 NRS unit after receiving a given dose vs. not. Based on this 38 per group are needed. Using the same dataset 52% of those in the active group improved by at least this amount. For a total sample of N, there are N/3 subjects who receive 0mg, 8mgand 16mg at week 1. In the control arm (0mg) there are no responses at the end of the first week. For the N/6 subjects receiving 8mg at the start of week 2, N/6*0.52 are expected to respond. In the arm receiving 8mg, N/3*0.52 are expected to respond at the end of the first week. Of the N/3*0 .48 that didn't respond in the first week 52% are expected to respond at the end of the second week. The same situation pertains to the group receiving 16mg at the start of week 1. For the sample of 135 subjects this implies that 82 in total are expected to respond. Assuming equal numbers are randomised to receiving the next incremental dose or remaining on the same dose this provides over 80% power.

Allowing for 20% attrition requires a total sample size of 171 subjects.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Physician diagnosed COPD confirmed by spirometry with the most recent result available defined as a prior post-bronchodilator FEV1/FVC < 0.7 in accordance with the GOLD 2014 criteria.
* Respiratory physician confirmed optimisation of treatment of COPD.
* On stable medications relating to the optimal treatment of COPD or its symptomatic management over the prior week except routine "as needed" medications.
* Breathlessness of a level three (3) or four (4) on the modified Medical Research Council (mMRC) breathlessness scale.
* worst breathlessness intensity in the previous 24 hours was at least 3/10 on a 0-10 numerical rating scale (NRS).
* English speaking with sufficient reading and writing ability to complete the study questionnaires
* Assessed as competent (using St Louise University Mental Status Examination (SLUMS) score of 27/30 for people whose highest level of education was high school, and 25/30 for people who did not complete high school).
* Able and willing to give written informed consent.

Exclusion Criteria:

* On any opioid for breathlessness in the previous seven (7) days.
* On regularly prescribed opioid medications for other conditions, including codeine preparations at or above 8mg oral morphine equivalent daily dose (MEDD) in the previous seven (7) days.
* History of adverse reactions to any of the study medications or constituents in the placebo;
* Australian-modified Karnofsky performance score (AKPS) less than 50 at the beginning of the study.
* Respiratory or cardiac event in the previous one week (excluding upper respiratory tract infections). Illness must have resolved completely prior to baseline evaluation, as judged by the person's treating physician.
* Evidence of respiratory depression with resting respiratory rate <8/min.
* Documented central hypoventilation syndrome.
* Current history of abuse of alcohol, or recent history of substance misuse.
* Uncontrolled nausea, vomiting or evidence of a gastrointestinal tract obstruction.
* Renal dysfunction with creatinine clearance calculated (MDRD) less than 20 mls/minute.
* Evidence of severe hepatic impairment defined as transaminases or bilirubin >4x normal (Excluding Gilbert's syndrome)
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Estimated)
Dates: Start 2016-08-08 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline worst breathlessness intensity over the previous 24 hours | Week 1
  Rated on a 0-10 numerical rating scale (NRS). Measured at baseline, Stage1-3 (daily diary) and Stage 4 (weekly diary). The primary endpoint is:
  * The difference between morphine sulphate 8mg and placebo (end of week1)
  * The difference of morphine sulphate 16 mg and placebo (end of week 1)
Change from the baseline in the number of steps per day | Week 3
  Difference from the baseline in the number of steps per day measured using the Fitbit(Charge HR). Measured at baseline, end of week 1, and end of week 3. The primary endpoint is:
  * The difference between morphine sulphate 8mg and placebo (end of week 1)
  * The difference between morphine sulphate 16mg and placebo (end of week 1)
  * Comparison between baseline and end of week 3

SECONDARY OUTCOMES:
Change from baseline end-tidal carbon dioxide | Up to week 15
  Measured at baseline and at the weekly visit for the randomisation phase, and then at the study exit in order to assess the theoretical risk of opioids worsening respiratory failure. Stages 1-4.
Change from baseline pulse oximetry | Up to week 15
  Measured at baseline and at the weekly visit for the randomisation phase, and then at the study exit in order to assess the theoretical risk of opioids worsening respiratory failure. Concomitant use of oxygen will be recorded. Stages 1-4.
Change from baseline intensity of breathlessness "average" | Up to week 15
  Rated on a 0-10 numerical rating scale (NRS). Measured at baseline, weeks 1-3 (daily diary) and stage 4 (weekly diary).
Change from baseline distress from breathlessness over the previous 24 hours | Up to week 15
  Rated on a 0-10 numerical rating scale (NRS). Measured at baseline, weeks 1-3 (daily diary) and stage 4 (weekly diary).
Change from baseline perceived-impact of breathlessness | Up to week 3
  Chronic Respiratory Questionnaire - Dyspnoea and Mastery Subscales. Baseline and end of Weeks 1-3.
Change from baseline functional impact of breathlessness | Up to week 15
  Rated on the Modified Medical Research Council Breathlessness Scale (mMRC). Measured at baseline and at the conclusion of the study.
Change from baseline sleep minutes | Week 3
  Measured using the Fitbit(Charge HR). Assessed at baseline (2 days), weeks 1 and 3.
Change from baseline sleep activity | Week 3
  Measured using the Fitbit(Charge HR). Given in number of movements per night (e.g. rolling over). Assessed at baseline (2 days), weeks 1 and 3.
Change from baseline in activity levels | Week 3
  Measured using the Fitbit(Charge HR). Difference from baseline in the number of active minutes per day. Assessed at baseline (2 days), weeks 1 and 3.
Change from baseline total energy expenditure | Week 3
  Measured using the Fitbit(Charge HR). Difference from baseline number of calories spent per day. Assessed at baseline (2 days), weeks 1 and 3.
Change from baseline performance status | Up to week 15
  Measured using Australian-modified Karnofsky Performance Status (AKPS). Baseline, Stage1, Stage2, Stage3 and Stage 4.
Change from baseline activities of daily living | Up to week 15
  Measured using Barthel Index. Baseline and Stage 4.
Change from baseline in sleep quality | Up to week 15
  Rated on a 4 point Likert scale. Measured at baseline, weeks 1-3 (daily diary) and stage 4 (weekly diary).
Change from baseline in objective sleep testing | Week 3
  Thirty (30) participants at the Sydney and Adelaide sites will be invited to undertake a simple, non-invasive home sleep study using the ResMed ApneaLink Plus device. Baseline and Stage3.
Change from baseline Polysomnography | Week 3
  Up to ten (10) participants will also undergo two (baseline and Stage 1) in-laboratory overnight sleep studies in Sydney and Adelaide.
Change from baseline Driving ability | Week 3 + 2 days
  Twenty (20) participants in Adelaide and Sydney. Baseline and on day 2 and 7 of the first week in an office-based simulator - AusEd.
Pharmacogenetic opioid profile - Number of participants with UGT2B7*2 and *28 polymorphisms | Baseline (1 day)
  The baseline blood samples will be analysed to detect the presence of UGT2B7*2 and *28 polymorphisms.
Pharmacogenetic opioid profile - Number of participants with P-glycoprotein polymorphism (ABCB1 5SNPs in a haplotype block) | Baseline (1 day)
  The baseline blood samples will be analysed to detect the presence of P-glycoprotein polymorphism (ABCB1 5SNPs in a haplotype block)
Pharmacogenetic opioid profile - Number of participants with 5-hydroxytryptamine type 3B (HTR3B) gene rs7103572 polymorphism | Baseline (1 day)
  The baseline blood samples will be analysed to detect the presence of 5-hydroxytryptamine type 3B (HTR3B) gene rs7103572 polymorphism
Pharmacogenetic opioid profile - Mu receptor (A118G) polymorphism | Baseline (1 day)
  The baseline blood samples will be analysed to detect the presence of Mu receptor (A118G) polymorphism
Pharmacokinetic (PK)/ Pharmacodynamic (PD) opioid profile: Morphine Peak Plasma Concentration [Cmax] | Week 1
  In a subset of 55 participants, morphine peak plasma concentrations will be analysed (4 blood samples over 8 hours) at steady state (end of week 1).
Pharmacokinetic (PK)/ Pharmacodynamic (PD) opioid profile: Morphine Area Under the Curve (AUC) | Week 1
  In a subset of 55 participants, morphine AUC will be analysed (4 blood samples over 8 hours) at steady state (end of week 1).
Pharmacokinetic (PK)/ Pharmacodynamic (PD) opioid profile: Morphine-6-glucuronide (M6G) Peak Plasma Concentration [Cmax] | Week 1
  In a subset of 55 participants, M6G Peak Plasma Concentration will be analysed (4 blood samples over 8 hours) at steady state (end of week 1).
Pharmacokinetic (PK)/ Pharmacodynamic (PD) opioid profile: Morphine-6-glucuronide (M6G) Area Under the Curve (AUC) | Week 1
  In a subset of 55 participants, M6G AUC will be analysed (4 blood samples over 8 hours) at steady state (end of week 1).
Pharmacokinetic (PK)/ Pharmacodynamic (PD) opioid profile: Morphine-3-glucuronide (M3G) Peak Plasma Concentration [Cmax] | Week 1
  In a subset of 55 participants, M3G Peak Plasma Concentration will be analysed (4 blood samples over 8 hours) at steady state (end of week 1).
Pharmacokinetic (PK)/ Pharmacodynamic (PD) opioid profile: Morphine-3-glucuronide (M3G) Area Under the Curve (AUC) | Week 1
  In a subset of 55 participants, M3G AUC will be analysed (4 blood samples over 8 hours) at steady state (end of week 1).
Change from baseline serum testosterone level | Week 15
  Baseline and study completion. To explore whether longer term morphine treatment is associated with decreased levels of testosterone.
Adverse Effects | Up to 15 weeks
  Rated on a Lickert Scale. Baseline, weeks 1-3 (daily diary), Stage 4 (weekly diary): Includes constipation, anxiety, appetite, nausea, vomiting, drowsiness, difficulty thinking clearly, problems passing urine, itch, other symptoms.
Change from baseline in concurrent symptoms | Up to 15 weeks
  Measured using the Edmonton Symptoms Assessment Scale (ESAS)
Change from the baseline anxiety and depression | Up to Week 15
  Rated using the Hospital Anxiety and Depression Scale (HADS). At baseline, completion of randomization stage and study exit.
Change in baseline global impression of change | Up to 15 weeks
  Participant-rated 7 point scale of the perception of their change, specifically their improvement since the commencement of the study. Measured at the end of Stages 1-3 and conclusion.
Change from baseline health-related quality of life | Up to 15 weeks
  Measured with EQ-5D-5L questionnaire. Baseline, Stages 1-3, Stage 4, conclusion.
Change from baseline health-status in COPD | Week 3
  Measured with the COPD Assessment Test (CAT) Baseline, Stages 1-3, Stage 4 and conclusion.
Blinded-patient preference to continue the treatment [3-point Likert Scale] | Up to week 15
  Asked at the end of week 1 and at the conclusion/drop-out of the study. A 3-point Likert scale will be used.
Change from baseline caregiver Impact | Up to week 15
  Scored using the Zarit Burden Interview (ZBI) 12 item short-form questionnaire. Baseline, end of weeks 1-3, stage 4.
Economic Evaluation - Cost per responder | Up to week 4
  From randomisation to 28 days post treatment or death (whichever is the shorter period). Estimated based on all health-care contacts including length of hospitalizations, emergency department visits, DRG codes, community health visits, GP and community nurse visits, outpatient visits and date of death. These participant level data allow within trial modeling using bootstrapping methods of replicates for costs and consequences of alternative strategies, allowing for covariance between costs and effects. Incremental net monetary benefit and cost-effectiveness acceptability curves will be estimated at potential threshold values for an additional responder.
Opioid Withdrawal | Up to week 15 + 3 days
  Evaluation using the Subjective Opioid Withdrawal Scale (SOWS) for 3 consecutive days. After the completion of the study (Weeks 1-15).

CONTACTS AND LOCATIONS:
Overall Officials: David C Currow, MD, PhD, Principal Investigator — Study Principal Investigator; Flinders University
Locations (15):
- Australia (14):
  - Clare Holland House, Canberra, Australian Capital Territory
  - Concord Hospital, Concord, New South Wales
  - St Vincent's Hospital Sydney - Sacred Heart Hospice, Darlinghurst, New South Wales
  - Calvary Health Care Kogarah, Kogarah, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Prince Charles Hospital, Brisbane, Queensland
  - Nambour Hospital, Sunshine Coast, Queensland
  - Southern Adelaide Palliative Services, Adelaide, South Australia
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Barwon Health McKellar Centre, Geelong, Victoria
  - The Austin Hospital, Heidelberg, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Perth, Western Australia
- Canterbury Respiratory Services, Christchurch, New Zealand

REFERENCES:
- [Derived] Ferreira DH, Ryan R, Smyth N, Clow A, Currow DC. The longitudinal impact of low-dose morphine on diurnal cortisol profiles in people with chronic breathlessness and chronic obstructive pulmonary disease (COPD): an exploratory study. Respir Res. 2025 Apr 23;26(1):156. doi: 10.1186/s12931-025-03230-9. PMID 40269943
- [Derived] Ekstrom M, Alameri F, Chang S, Ferreira D, Johnson MJ, Currow DC. Harms of Morphine for Chronic Breathlessness in Relation to Dose, Duration and Titration Phase. J Pain Symptom Manage. 2025 Jun;69(6):581-588.e2. doi: 10.1016/j.jpainsymman.2025.02.020. Epub 2025 Feb 25. PMID 40015533
- [Derived] Altree TJ, Toson B, Loffler KA, Ekstrom M, Currow DC, Eckert DJ. Low-Dose Morphine Does Not Cause Sleepiness in Chronic Obstructive Pulmonary Disease: A Secondary Analysis of a Randomized Clinical Trial. Am J Respir Crit Care Med. 2024 Nov 1;210(9):1113-1122. doi: 10.1164/rccm.202310-1780OC. PMID 38477675
- [Derived] Ekstrom M, Ferreira D, Chang S, Louw S, Johnson MJ, Eckert DJ, Fazekas B, Clark KJ, Agar MR, Currow DC; Australian National Palliative Care Clinical Studies Collaborative. Effect of Regular, Low-Dose, Extended-release Morphine on Chronic Breathlessness in Chronic Obstructive Pulmonary Disease: The BEAMS Randomized Clinical Trial. JAMA. 2022 Nov 22;328(20):2022-2032. doi: 10.1001/jama.2022.20206. PMID 36413230
- [Derived] Ferreira DH, Kochovska S, Honson A, Phillips JL, Currow DC. Two faces of the same coin: a qualitative study of patients' and carers' coexistence with chronic breathlessness associated with chronic obstructive pulmonary disease (COPD). BMC Palliat Care. 2020 May 6;19(1):64. doi: 10.1186/s12904-020-00572-7. PMID 32375747
- [Derived] Currow D, Watts GJ, Johnson M, McDonald CF, Miners JO, Somogyi AA, Denehy L, McCaffrey N, Eckert DJ, McCloud P, Louw S, Lam L, Greene A, Fazekas B, Clark KC, Fong K, Agar MR, Joshi R, Kilbreath S, Ferreira D, Ekstrom M; Australian national Palliative Care Clinical Studies Collaborative (PaCCSC). A pragmatic, phase III, multisite, double-blind, placebo-controlled, parallel-arm, dose increment randomised trial of regular, low-dose extended-release morphine for chronic breathlessness: Breathlessness, Exertion And Morphine Sulfate (BEAMS) study protocol. BMJ Open. 2017 Jul 17;7(7):e018100. doi: 10.1136/bmjopen-2017-018100. PMID 28716797